CLINICAL TRIAL: NCT02146482
Title: Evaluating Change in Back Pain From Access to a Sit-stand Workstation
Brief Title: Access to a Sit-stand Computer Workstation and Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kathleen Horst, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSCWStanford
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Results first posted 2015-06-19 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Low Back Pain; Back Pain
Keywords: back pain; low back pain; sit-stand workstation; standing desk
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Did not receive an intervention during the active portion of the study (i.e. 12 weeks). After the active portion of the study, this group was given a sit-stand computer workstation.
- Sit-stand computer workstation (Experimental): Given a sit-stand computer workstation to use at their place of work
  Interventions: Other: Sit-stand computer workstation

INTERVENTIONS:
Other: Sit-stand computer workstation — A sit-stand computer workstation allows one to sit or stand throughout the day while maintaining continued use of one's computer.
  Other Names: Standing desk; WorkFit
  Arms: Sit-stand computer workstation

SUMMARY:
The purpose of the study is to evaluate the changes in back pain from access to a sit-stand workstation. Other muscle and joint pain and/or discomfort will also be evaluated. We hypothesize that access to a sit-stand workstation will allow one to experience postural variation and reduce back pain.

ELIGIBILITY:
Inclusion Criteria:

* Back pain lasting ≥3 months and reported at a minimum of 4 out of 10 on the pain scale.
* Sits >6 hours out of an 8-hour work day for work purposes
* Able and willing to fill out a daily survey for the first week prior to randomization
* Participants must be >18 years of age. There are no gender/race-ethnic restrictions.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Unable to stand for at least 10 minutes.
* Currently using a sit-stand desk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen C Horst, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Background] Woolf AD, Pfleger B. Burden of major musculoskeletal conditions. Bull World Health Organ. 2003;81(9):646-56. Epub 2003 Nov 14. PMID 14710506
- [Background] Martin BI, Deyo RA, Mirza SK, Turner JA, Comstock BA, Hollingworth W, Sullivan SD. Expenditures and health status among adults with back and neck problems. JAMA. 2008 Feb 13;299(6):656-64. doi: 10.1001/jama.299.6.656. PMID 18270354
- [Background] Hamilton MT, Healy GN, Dunstan DW, Zderic TW, Owen N. Too Little Exercise and Too Much Sitting: Inactivity Physiology and the Need for New Recommendations on Sedentary Behavior. Curr Cardiovasc Risk Rep. 2008 Jul;2(4):292-298. doi: 10.1007/s12170-008-0054-8. PMID 22905272
- [Background] Morl F, Bradl I. Lumbar posture and muscular activity while sitting during office work. J Electromyogr Kinesiol. 2013 Apr;23(2):362-8. doi: 10.1016/j.jelekin.2012.10.002. Epub 2012 Nov 2. PMID 23122693
- [Background] Hamburg NM, McMackin CJ, Huang AL, Shenouda SM, Widlansky ME, Schulz E, Gokce N, Ruderman NB, Keaney JF Jr, Vita JA. Physical inactivity rapidly induces insulin resistance and microvascular dysfunction in healthy volunteers. Arterioscler Thromb Vasc Biol. 2007 Dec;27(12):2650-6. doi: 10.1161/ATVBAHA.107.153288. Epub 2007 Oct 11. PMID 17932315
- [Background] Ekblom-Bak E, Hellenius ML, Ekblom O, Engstrom LM, Ekblom B. Independent associations of physical activity and cardiovascular fitness with cardiovascular risk in adults. Eur J Cardiovasc Prev Rehabil. 2010 Apr;17(2):175-80. doi: 10.1097/HJR.0b013e32833254f2. PMID 19809331
- [Background] Zderic TW, Hamilton MT. Physical inactivity amplifies the sensitivity of skeletal muscle to the lipid-induced downregulation of lipoprotein lipase activity. J Appl Physiol (1985). 2006 Jan;100(1):249-57. doi: 10.1152/japplphysiol.00925.2005. Epub 2005 Sep 29. PMID 16195388
- [Background] Katzmarzyk PT, Church TS, Craig CL, Bouchard C. Sitting time and mortality from all causes, cardiovascular disease, and cancer. Med Sci Sports Exerc. 2009 May;41(5):998-1005. doi: 10.1249/MSS.0b013e3181930355. PMID 19346988
- [Background] Pedersen BK. The diseasome of physical inactivity--and the role of myokines in muscle--fat cross talk. J Physiol. 2009 Dec 1;587(Pt 23):5559-68. doi: 10.1113/jphysiol.2009.179515. Epub 2009 Sep 14. PMID 19752112
- [Background] Pedersen BK. Muscles and their myokines. J Exp Biol. 2011 Jan 15;214(Pt 2):337-46. doi: 10.1242/jeb.048074. PMID 21177953
- [Background] Pillastrini P, Mugnai R, Bertozzi L, Costi S, Curti S, Guccione A, Mattioli S, Violante FS. Effectiveness of an ergonomic intervention on work-related posture and low back pain in video display terminal operators: a 3 year cross-over trial. Appl Ergon. 2010 May;41(3):436-43. doi: 10.1016/j.apergo.2009.09.008. Epub 2009 Oct 23. PMID 19853837
- [Background] IJmker S, Huysmans MA, Blatter BM, van der Beek AJ, van Mechelen W, Bongers PM. Should office workers spend fewer hours at their computer? A systematic review of the literature. Occup Environ Med. 2007 Apr;64(4):211-22. doi: 10.1136/oem.2006.026468. Epub 2006 Nov 9. PMID 17095550
- [Background] Robertson M, Amick BC 3rd, DeRango K, Rooney T, Bazzani L, Harrist R, Moore A. The effects of an office ergonomics training and chair intervention on worker knowledge, behavior and musculoskeletal risk. Appl Ergon. 2009 Jan;40(1):124-35. doi: 10.1016/j.apergo.2007.12.009. Epub 2008 Mar 11. PMID 18336791
- [Background] Amick BC 3rd, Robertson MM, DeRango K, Bazzani L, Moore A, Rooney T, Harrist R. Effect of office ergonomics intervention on reducing musculoskeletal symptoms. Spine (Phila Pa 1976). 2003 Dec 15;28(24):2706-11. doi: 10.1097/01.BRS.0000099740.87791.F7. PMID 14673374
- [Background] Aaras A, Horgen G, Bjorset HH, Ro O, Walsoe H. Musculoskeletal, visual and psychosocial stress in VDU operators before and after multidisciplinary ergonomic interventions. A 6 years prospective study--Part II. Appl Ergon. 2001 Dec;32(6):559-71. doi: 10.1016/s0003-6870(01)00030-8. PMID 11703042
- [Background] Hakala PT, Rimpela AH, Saarni LA, Salminen JJ. Frequent computer-related activities increase the risk of neck-shoulder and low back pain in adolescents. Eur J Public Health. 2006 Oct;16(5):536-41. doi: 10.1093/eurpub/ckl025. Epub 2006 Mar 8. PMID 16524936
- [Background] Andersson GB. Epidemiologic aspects on low-back pain in industry. Spine (Phila Pa 1976). 1981 Jan-Feb;6(1):53-60. doi: 10.1097/00007632-198101000-00013. PMID 6451937
- [Background] Videman T, Nurminen M, Troup JD. 1990 Volvo Award in clinical sciences. Lumbar spinal pathology in cadaveric material in relation to history of back pain, occupation, and physical loading. Spine (Phila Pa 1976). 1990 Aug;15(8):728-40. PMID 2146754
- [Background] Frymoyer JW, Pope MH, Costanza MC, Rosen JC, Goggin JE, Wilder DG. Epidemiologic studies of low-back pain. Spine (Phila Pa 1976). 1980 Sep-Oct;5(5):419-23. doi: 10.1097/00007632-198009000-00005. PMID 6450452
- [Background] Nakazawa T, Okubo Y, Suwazono Y, Kobayashi E, Komine S, Kato N, Nogawa K. Association between duration of daily VDT use and subjective symptoms. Am J Ind Med. 2002 Nov;42(5):421-6. doi: 10.1002/ajim.10133. PMID 12382255
- [Background] Fogleman M, Lewis RJ. Factors associated with self-reported musculoskeletal discomfort in video display terminal (VDT) users. Int J Ind Ergonom 29(6):311-8, 2002.
- [Background] Hartvigsen J, Kyvik KO, Leboeuf-Yde C, Lings S, Bakketeig L. Ambiguous relation between physical workload and low back pain: a twin control study. Occup Environ Med. 2003 Feb;60(2):109-14. doi: 10.1136/oem.60.2.109. PMID 12554838
- [Background] Roffey DM, Wai EK, Bishop P, Kwon BK, Dagenais S. Causal assessment of occupational sitting and low back pain: results of a systematic review. Spine J. 2010 Mar;10(3):252-61. doi: 10.1016/j.spinee.2009.12.005. Epub 2010 Jan 25. PMID 20097618
- [Background] Dugan SA. The role of exercise in the prevention and management of acute low back pain. Clin Occup Environ Med. 2006;5(3):615-32, vi-vii. doi: 10.1016/j.coem.2006.03.003. PMID 16963378
- [Background] Katz JN. Lumbar disc disorders and low-back pain: socioeconomic factors and consequences. J Bone Joint Surg Am. 2006 Apr;88 Suppl 2:21-4. doi: 10.2106/JBJS.E.01273. PMID 16595438
- [Background] Hwang JA, Bae SH, Do Kim G, Kim KY. The effects of sensorimotor training on anticipatory postural adjustment of the trunk in chronic low back pain patients. J Phys Ther Sci. 2013 Sep;25(9):1189-92. doi: 10.1589/jpts.25.1189. Epub 2013 Oct 20. PMID 24259943
- [Background] Zemp R, Taylor WR, Lorenzetti S. In vivo spinal posture during upright and reclined sitting in an office chair. Biomed Res Int. 2013;2013:916045. doi: 10.1155/2013/916045. Epub 2013 Sep 24. PMID 24175307
- [Background] Lee SH, Kim TH, Lee BH. The effect of abdominal bracing in combination with low extremity movements on changes in thickness of abdominal muscles and lumbar strength for low back pain. J Phys Ther Sci. 2014 Jan;26(1):157-60. doi: 10.1589/jpts.26.157. Epub 2014 Feb 6. PMID 24567697
- [Background] Lee CW, Hwangbo K, Lee IS. The effects of combination patterns of proprioceptive neuromuscular facilitation and ball exercise on pain and muscle activity of chronic low back pain patients. J Phys Ther Sci. 2014 Jan;26(1):93-6. doi: 10.1589/jpts.26.93. Epub 2014 Feb 6. PMID 24567683
- [Background] Tekur P, Nagarathna R, Chametcha S, Hankey A, Nagendra HR. A comprehensive yoga programs improves pain, anxiety and depression in chronic low back pain patients more than exercise: an RCT. Complement Ther Med. 2012 Jun;20(3):107-18. doi: 10.1016/j.ctim.2011.12.009. Epub 2012 Jan 28. PMID 22500659
- [Background] Pinto RZ, Ferreira PH, Kongsted A, Ferreira ML, Maher CG, Kent P. Self-reported moderate-to-vigorous leisure time physical activity predicts less pain and disability over 12 months in chronic and persistent low back pain. Eur J Pain. 2014 Sep;18(8):1190-8. doi: 10.1002/j.1532-2149.2014.00468.x. Epub 2014 Feb 27. PMID 24577780
- [Background] Yoo WG. Effect of Resting in a Chair, Resting with Range of Motion Exercises, and Back Strengthening Exercises on Pain and the Flexion-relaxation Ratio of Computer Workers with Low Back Pain. J Phys Ther Sci. 2014 Feb;26(2):321-2. doi: 10.1589/jpts.26.321. Epub 2014 Feb 28. PMID 24648658
- [Background] Schiphorst Preuper HR, Geertzen JH, van Wijhe M, Boonstra AM, Molmans BH, Dijkstra PU, Reneman MF. Do analgesics improve functioning in patients with chronic low back pain? An explorative triple-blinded RCT. Eur Spine J. 2014 Apr;23(4):800-6. doi: 10.1007/s00586-014-3229-7. Epub 2014 Feb 15. PMID 24526247
- [Background] Ebadi S, Henschke N, Nakhostin Ansari N, Fallah E, van Tulder MW. Therapeutic ultrasound for chronic low-back pain. Cochrane Database Syst Rev. 2014 Mar 14;(3):CD009169. doi: 10.1002/14651858.CD009169.pub2. PMID 24627326
- [Background] Hartvigsen J, Leboeuf-Yde C, Lings S, Corder EH. Is sitting-while-at-work associated with low back pain? A systematic, critical literature review. Scand J Public Health. 2000 Sep;28(3):230-9. PMID 11045756
- [Background] Keller S, Bann CM, Dodd SL, Schein J, Mendoza TR, Cleeland CS. Validity of the brief pain inventory for use in documenting the outcomes of patients with noncancer pain. Clin J Pain. 2004 Sep-Oct;20(5):309-18. doi: 10.1097/00002508-200409000-00005. PMID 15322437
- [Background] Roland M, Morris R. A study of the natural history of back pain. Part I: development of a reliable and sensitive measure of disability in low-back pain. Spine (Phila Pa 1976). 1983 Mar;8(2):141-4. doi: 10.1097/00007632-198303000-00004. No abstract available. PMID 6222486
- [Background] Husemann B, Von Mach CY, Borsotto D, Zepf KI, Scharnbacher J. Comparisons of musculoskeletal complaints and data entry between a sitting and a sit-stand workstation paradigm. Hum Factors. 2009 Jun;51(3):310-20. doi: 10.1177/0018720809338173. PMID 19750794
- [Background] Tissot F, Messing K, Stock S. Studying the relationship between low back pain and working postures among those who stand and those who sit most of the working day. Ergonomics. 2009 Nov;52(11):1402-18. doi: 10.1080/00140130903141204. PMID 19851907
- [Background] Benden ME, Blake JJ, Wendel ML, Huber JC Jr. The impact of stand-biased desks in classrooms on calorie expenditure in children. Am J Public Health. 2011 Aug;101(8):1433-6. doi: 10.2105/AJPH.2010.300072. Epub 2011 Mar 18. PMID 21421945
- [Background] Reiff C, Marlatt K, Dengel DR. Difference in caloric expenditure in sitting versus standing desks. J Phys Act Health. 2012 Sep;9(7):1009-11. doi: 10.1123/jpah.9.7.1009. PMID 22971879
- [Background] Healy GN, Dunstan DW, Salmon J, Cerin E, Shaw JE, Zimmet PZ, Owen N. Breaks in sedentary time: beneficial associations with metabolic risk. Diabetes Care. 2008 Apr;31(4):661-6. doi: 10.2337/dc07-2046. Epub 2008 Feb 5. PMID 18252901
- [Background] Healy GN, Dunstan DW, Salmon J, Cerin E, Shaw JE, Zimmet PZ, Owen N. Objectively measured light-intensity physical activity is independently associated with 2-h plasma glucose. Diabetes Care. 2007 Jun;30(6):1384-9. doi: 10.2337/dc07-0114. Epub 2007 May 1. PMID 17473059
- [Background] Owen N, Healy GN, Matthews CE, Dunstan DW. Too much sitting: the population health science of sedentary behavior. Exerc Sport Sci Rev. 2010 Jul;38(3):105-13. doi: 10.1097/JES.0b013e3181e373a2. PMID 20577058
- [Background] Krause N, Lynch JW, Kaplan GA, Cohen RD, Salonen R, Salonen JT. Standing at work and progression of carotid atherosclerosis. Scand J Work Environ Health. 2000 Jun;26(3):227-36. doi: 10.5271/sjweh.536. PMID 10901115

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Sit-stand Computer Workstation
Started | 21 (11 participants total enrolled in study but withdrew prior to randomization) | 25 (11 participants total enrolled in study but withdrew prior to randomization)
Completed | 21 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Sit-stand Computer Workstation | Total
Number analyzed (Participants) | 21 | 25 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 25 | 46
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 21 | 25 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change in Back Pain
Description: The Roland-Morris Disability Questionnaire is designed to assess self-rated physical disability caused by low back pain. The patient is asked to agree or disagree with 24 different statements related to their back pain. The end score is the sum of the agreed statements. The score ranges from 0 (no disability) to 24 (maximum disability).
Time Frame: Baseline (Week 1) and Follow-Up (Week 18)
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Control | Sit-stand Computer Workstation
Number analyzed (Participants) | 21 | 25
units on a scale
  Baseline | 6 [0 to 15] | 8.5 [1 to 15]
  Follow Up | 4 [0 to 12] | 1.5 [0 to 19]

2. Secondary Outcome: Change in Pain in Other Body Parts
Description: The Brief Pain Inventory (BPI) allows patients to rate the severity of their pain and the degree to which their pain interferes with common dimensions of feeling and function. This data was not analyzed due to the focus of the project on lower back pain.
Time Frame: At the conclusion of each work day for 12 weeks and 8 weeks later
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Control | Sit-stand Computer Workstation
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/25
Other Adverse Events (participants affected / at risk) | 0/21 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No